CLINICAL TRIAL: NCT06922474
Title: Molecular Epidemiology of Enteroviruses Detected at the Virology Laboratory of Brest University Hospital During the Period 2018-2024: Retrospective Analysis of an Atypical Meningitis Epidemic in 2024
Brief Title: Molecular Epidemiology of Enteroviruses Detected at the Virology Laboratory of Brest University Hospital During the Period 2018-2024: Retrospective Analysis of an Atypical Meningitis Epidemic in 2024 (BrEcho9Men)
Acronym: BrEcho9Men
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC25.0054 - BrEcho9Men
Record Dates: First submitted 2025-04-03; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-03

CONDITIONS: Enterovirus Infections; Meningitis, Viral; Meningitis Enterovirus; Echovirus 9
Keywords: Echovirus 9; Enterovirus; Viral meningitis; Molecular epidemiology; Phylogenetic analysis; RT-PCR; Retrospective study; Surveillance; France; outbreak; Emerging variant; France epidemiology
MeSH Terms: conditions — Enterovirus Infections; Meningitis, Viral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Clinical specimens tested positive for enteroviruses by RT-PCR will be retained. These include cerebrospinal fluid (CSF), throat swabs, stool samples, and nasopharyngeal swabs collected as part of routine care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is being done to learn more about enterovirus infections detected in the cerebrospinal fluid of patients at CHU de Brest. Researchers will analyze medical records and laboratory data collected between 2018 and 2024. They will look at how these infections present in patients, and whether a specific virus type, called Echo-9, may be associated with different clinical features or represent an emerging variant.

ELIGIBILITY:
Inclusion Criteria:

* Cerebrospinal fluid (CSF) sample positive for enterovirus by RT-PCR between January 1, 2018 and December 31, 2024 , performed at the virology laboratory of CHU de Brest.
* No documented opposition to the use of medical data for research purposes.

Exclusion Criteria:

* Patients under legal protection (guardianship, curatorship, etc.)
* Refusal to participate in the study

Ages: 0 Days to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a cerebrospinal fluid sample positive for enterovirus by RT-PCR performed at the virology laboratory of CHU de Brest between 2018 and 2024. This includes patients managed at CHU de Brest as well as at partner hospitals in Finistère (France) whose samples were processed centrally.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Phylogenetic analysis of Echo-9 strains detected between 2018 and 2024 | January 1, 2018 to December 31, 2024
  Molecular characterization and phylogenetic comparison of Echo-9 strains detected at CHU de Brest and throughout France between January 1, 2018 and December 31, 2024, to identify a possible emerging variant.

SECONDARY OUTCOMES:
Temporal distribution of enterovirus infections documented at CHU de Brest | January 1, 2018 to December 31, 2024
  Weekly quantification of enterovirus-positive cases (by RT-PCR) detected at CHU de Brest from 2018 to 2024. Comparison with national surveillance data from the French National Reference Center to detect atypical epidemic peaks, with a focus on 2024.
Clinical characteristics of enterovirus-positive CSF cases | January 1, 2018 to December 31, 2024
  Among patients with cerebrospinal fluid samples positive for enterovirus between 2018 and 2024, clinical features will be described, including headache intensity, clinical severity, infection site (CSF, throat, stool, nasopharyngeal samples), and use of morphine. Subgroup comparisons may be conducted according to enterovirus genotype and year of infection, depending on the results of molecular typing.
Biological characteristics of enterovirus-positive CSF samples | January 1, 2018 to December 31, 2024
  Among patients with cerebrospinal fluid samples positive for enterovirus between 2018 and 2024, biological parameters from positive samples will be described. For cerebrospinal fluid samples, variables include white blood cell count with differential, protein level, and the cerebrospinal fluid to blood glucose ratio. The presence or absence of additional positive samples (throat, stool, nasopharyngeal swabs) will also be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement